CLINICAL TRIAL: NCT02263586
Title: Acid-base and Electrolyte Balance Among Triathletes in the Ironman European Championship
Brief Title: Influence of Triathlon on the Electrolyte Balance
Acronym: Ironman
Status: Completed | Type: Observational
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Dr. med. Stefan Braunecker, Anesthesiologist, Researcher, University Hospital of Cologne
Other Study IDs: Ironman
Record Dates: First submitted 2014-10-04; First posted 2014-10-13 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Hyponatremia
Keywords: Ironman; Triathlon
MeSH Terms: conditions — Hyponatremia | interventions — Educational Status; Nutritional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Education in nutrition — Athletes were given a 45 min lesson on the proper diet and fluid intake to prevent hyponatremia in long-distance triathlon.

SUMMARY:
Aim of the study is examining the incidence of the occurrence of hyponatremia during a Triathlon

DETAILED DESCRIPTION:
Studies in similar endurance sports (e.g. marathon) could already indicate a high incidence for the appearance of hyponatremia during competitions. The loss of sodium through sweating and the excessive fluid intake during the competitions is a primary risk factor for the development of hyponatremia.

Based on the known occurrence of hyponatremia in marathon runners, participants of the Ironman European Championship between the years 2005 and 2014 were screened for the occurrence of hyponatremia after finishing the race for safety reasons. Subjects were approached at random in the athlete's garden and invited to participate. All participants were 18 years or older.

ELIGIBILITY:
Inclusion Criteria:

* finisher of a long-distance triathlon
* > 18 years
* < 60 years

Exclusion Criteria:

* not finished a long-distance triathlon
* < 18 years
* > 60 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants of a long-distance triathlon
Sampling Method: Probability Sample
Enrollment: 1089 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Electrolyte balance Blood sodium | within 20 minutes after finishing the race

SECONDARY OUTCOMES:
Acid balance | within 20 minutes after finishing the race

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Braunecker, M.D., Principal Investigator — University Hospital Cologne
Locations (1):
- Uniklinik Köln, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Almond CS, Shin AY, Fortescue EB, Mannix RC, Wypij D, Binstadt BA, Duncan CN, Olson DP, Salerno AE, Newburger JW, Greenes DS. Hyponatremia among runners in the Boston Marathon. N Engl J Med. 2005 Apr 14;352(15):1550-6. doi: 10.1056/NEJMoa043901. PMID 15829535